CLINICAL TRIAL: NCT04195139
Title: A Randomised Phase II Study of NivolUmab and TeMozolomide vs Temozolomide Alone in Newly Diagnosed Elderly Patients With Glioblastoma (NUTMEG)
Brief Title: Nivolumab and Temozolomide Versus Temozolomide Alone in Newly Diagnosed Elderly Patients With GBM
Acronym: NUTMEG
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sydney (Other)
Collaborators: Cooperative Trials Group for Neuro-Oncology (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COGNO 16/01, CTC 0156; ACTRN12617000267358 (Registry Identifier: Australian New Zealand Clinical Trials Registry)
Record Dates: First submitted 2019-11-18; First posted 2019-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Glioblastoma Multiforme
Keywords: GBM; Astrocytoma WHO grade IV; Elderly; Nivolumab; Temozolomide
MeSH Terms: conditions — Glioblastoma | interventions — Nivolumab; Temozolomide

STUDY DESIGN:
Intervention Model Description: All participants will receive radiotherapy (weekdays over 21 days) concurrently with temozolomide (TMZ) tablets 75mg/m2 daily for 21 days.
  After a 4 week break, participants will receive either experimental or standard treatment.
  Experimental treatment: Participants assigned to this group will receive nivolumab intravenous infusions (days 1 and 15 every 28 days with concurrent adjuvant temozolomide tablets days 1-5, every 28 days) for 6 cycles.
  Standard treatment: Participants assigned to this group will receive the standard treatment of adjuvant temozolomide (days 1-5 every 28 days) for 6 cycles.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nivolumab and Temozolomide (Experimental): After radiotherapy and 4 week break, participants who are assigned to this arm will receive Nivolumab with concurrent adjuvant temozolomide treatment
  Interventions: Drug: Nivolumab; Drug: Temozolomide
- Temozolomide (Active Comparator): After radiotherapy and 4 week break, participants who are assigned to this arm will receive the standard treatment of adjuvant temozolomide treatment
  Interventions: Drug: Temozolomide

INTERVENTIONS:
Drug: Nivolumab — Participants will receive Nivolumab intravenous infusions (240 mg days 1 and 15 every 28 days for cycles 1-4; then 480 mg day 1 every 28 days for cycles 5-6).
  Other Names: Opdivo
  Arms: Nivolumab and Temozolomide
Drug: Temozolomide — Participants will receive temozolomide (TMZ) tablets days 1-5, every 28 days for 6 cycles. TMZ will be dosed at 150mg/m2 for the first cycle. If well tolerated TMZ is then given at 200mg/m2 for cycles 2 - 6.
  Other Names: Temodar; Temodal; Temcad

SUMMARY:
This study aims to investigate effect of Nivolumab and Temozolomide vs Temozolomide alone on overall survival in newly diagnosed elderly patients with glioblastoma.

Who is it for? You may be eligible to join this study if you are aged 65 years or above, with newly diagnosed histologically confirmed GBM (WHO grade IV glioma including gliosarcoma) following surgery.

The study aims to evaluate whether the combination of adjuvant nivolumab with temozolomide improves overall survival outcomes for this patient population. The outcome of the study will help determine the most effective treatment for patients with glioblastoma in the future.

DETAILED DESCRIPTION:
Study details:

Participants will be allocated to either experimental or control group in a 2:1 ratio by chance (randomly). Patients assigned to the experimental group will receive a course of nivolumab via intravenous infusion (240 mg on days 1 and 15 every 28 days for cycles 1-4; then 480 mg day 1 every 28 days for cycles 5-6) in addition to the standard regimen of Temozolomide (TMZ) tablets and radiotherapy. Patients assigned to the control group will receive the standard treatment of adjuvant temozolomide (150-200mg/m2 days 1-5 every 28 days) for 6 cycles and standard radiotherapy treatment (40 Gy administered in 15 fractions).

ELIGIBILITY:
Inclusion Criteria:

1. Adults, aged greater than or equal to 70 years, or aged 65-69 years if long course RT is inappropriate, with newly diagnosed histologically confirmed GBM (WHO grade IV glioma including gliosarcoma) following surgery
2. Tissue available for MGMT testing
3. ECOG 0-2
4. Life expectancy of >12 weeks
5. Adequate bone marrow function (platelets > 100 x 10^9/L, ANC > 1.5 x 10^9/L)
6. Adequate liver function (ALT/AST < 1.5 x ULN)
7. Adequate renal function (creatinine clearance > 30 ml/min measured using Cockcroft-Gault
8. Willing and able to comply with all study requirements, including treatment, timing and/or nature of required assessments including MRI
9. Signed, written informed consent

Exclusion Criteria:

1. Specific comorbidities or conditions (e.g. psychiatric) or concomitant medications which may impact with the administration of study related treatments or procedures
2. Other co-morbidities or conditions that may compromise assessment of key outcomes
3. Prior chemotherapy or cranial radiation within the last 5 years. Prior or concomitant therapies for GBM (except surgery).
4. History of another malignancy within 2 years prior to registration. Patients with a past history of adequately treated carcinoma-in-situ, basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or superficial transitional cell carcinoma of the bladder are eligible. Patients with a history of other malignancies are eligible if they have been continuously disease free for at least 2 years after definitive primary treatment.
5. Significant infection, including chronic active hepatitis B, hepatitis C, or HIV. Testing for these is not mandatory unless clinically indicated
6. Active, known or suspected autoimmune disease. Subjects with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
7. For symptoms related to GBM, the need for >4 mg/day of dexamethasone or >20 mg/day prednisone (or equivalent) at the time of screening.
8. For a condition other than GBM, the need for >2 mg/day of dexamethasone or >10 mg/day prednisone (or equivalent) or other immunosuppressive medications within 14 days prior to randomisation. Exceptions to this include the use of inhaled or topical steroids >10 mg/day prednisone (or equivalent), which are permitted in the absence of active autoimmune disease.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 103 (Actual)
Dates: Start 2018-02-22 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival outcomes | 24 months post randomisation of first participant
  Overall survival is defined as the interval from the date of randomisation to date of death from any cause, or date of last known follow-up alive. This will be calculated using the Kaplan-Meier method.

SECONDARY OUTCOMES:
Progression Free Survival | 6 months post randomisation
  Progression free survival (PFS) is defined as the interval from date of randomisation to the date of first evidence of disease progression or death from any cause, whichever occurs first. The PFS will be calculated using the Kaplan-Meier method and disease progression is defined according to modified Response Assessment in Neuro-Oncology (RANO) criteria.
Number and severity of adverse events | Through study completion, up to 24 months
  The NCI Common Terminology Criteria for Adverse Events version 4.03 (NCI CTCAE v4.03) will be used to classify and grade the intensity of adverse events.
Health related quality of life of participants (QLQ C-30) | Through study completion, up to 24 months
  Health related quality of life will be reported directly by the participants using the EORTC core quality of life questionnaire QLQ C-30. The QLQ-C30 is a 30-item questionnaire with 5 functional scales (physical, role, cognitive, emotional, and social), global health status, 3 symptom scales (fatigue, pain, nausea/vomiting), and other (dyspnoea, appetite loss, insomnia, constipation/diarrhea, and financial difficulties). Most questions used 4-point scale (1 'Not at All' to 4 'Very Much'); 2 questions used 7-point scale (1 'Very Poor' to 7 'Excellent'). Scores are averaged and transformed to 0-100 scale; higher score=better level of physical functioning.
Health related quality of life of participants (QLQ-BN20) | Through study completion, up to 24 months
  Health related quality of life will be reported directly by the participants using the EORTC core quality of life questionnaire brain cancer specific module (QLQ-BN20). The QLQ-BN20 consisted of 20 items assessing visual disorders, motor dysfunction, communication deficit, various disease symptoms (e.g. headaches and seizures), treatment toxicities (e.g. hair loss) and future uncertainty. All of the 20 items are rated on a 4 point scale (1=not at all, 4=very much), and were linearly transformed to a 0-100 scale, with higher scores indicating more severe symptoms.
Health related quality of life of participants (EuroQoL EQ-5D-5L) | Through study completion, up to 24 months
  Health related quality of life will be reported directly by the participants using the EORTC core quality of life questionnaire EuroQol EQ-5D-5L. The EQ-5D-5L descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression and as overall health using a "thermometer" visual analog scale with response options ranging from 0 (worst imaginable health) to 100 (best imaginable health).
Neurologic function of participants | Through study completion, up to 24 months
  Cognitive function will be assessed by the Neurologic Assessment in Neuro-Oncology (NANO) scales. The NANO is a quantifiable evaluation of nine major domains for subjects with brain tumours. The domains include: gait, strength, ataxia, sensation, visual field, facial strength, language, level of consciousness, behaviour and overall. Each domain is rated on a scale of 0 to 3 where 0 represents normal and 3 represents the worst severity. The evaluation is based on direct observation/testing performed during routine office visits.
Correlating modified RANO and immune related RANO in the experimental arm | Through study completion, up to 24 months
  Site investigators will assess disease progression using modified RANO criteria for clinical decision making. The study team will coordinate image analysis and central review of MRI including modified RANO (both experimental and comparator arms) and iRANO (in the experimental arm).

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Khasraw, Study Chair — Duke University
Locations (20):
- Duke University Medical Center, Durham, North Carolina, United States
- Australia (19):
  - Campbelltown Hospital, Campbelltown, New South Wales
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Gosford Hospital, Gosford, New South Wales
  - Newcastle Private Hospital, New Lambton Heights, New South Wales
  - Port Macquarie Hospital, Port Macquarie, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Royal North Shore Hospital, Saint Leonards, New South Wales
  - Wollongong Hospital, Wollongong, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Icon Cancer Centre, South Brisbane, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Monash Medical Centre, Clayton, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Epworth Healthcare, Richmond, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Melo SM, Elias Nunes da Silva ME, Torloni MR, Riera R, De Cicco K, Latorraca CO, Pinto ACPN. Anti-PD-1 and anti-PD-L1 antibodies for glioma. Cochrane Database Syst Rev. 2025 Jan 8;1(1):CD012532. doi: 10.1002/14651858.CD012532.pub2. PMID 39777725